CLINICAL TRIAL: NCT05216237
Title: An Open-Label, Multi-Center, Phase II Study to Evaluate the Efficacy and Safety of PD-1 Antibody Sintilimab Plus Apatinib and Chemotherapy in Patients With HER-2 Negative MSS Advanced or Metastatic GC or GEJ Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of Sintilimab Plus Apatinib and Chemotherapy in Patients With HER-2 Negative Microsatellite Stability (MSS) Advanced or Metastatic Gastric (GC) or Gastroesophageal Junction (GEJ) Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiuda Zhao (Other)
Collaborators: Lanzhou University Second Hospital (Other)
Responsible Party: Sponsor-Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Organization: Affiliated Hospital of Qinghai University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHQU-2022001
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Gastric Cancer; Chemotherapy; Immunotherapy
Keywords: Gastric Cancer; Chemotherapy; Immunotherapy; Microsatellite stability
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; apatinib; BID protein, human; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Patients who meet the inclusion criteria will receive with sintilimab combined with apatinib and chemotherapy(Oxaliplatin plus Tegafur gimeracil oteracil potassium capsules). At the same time, tumor samples were collected for tissue PD-L1 detection and blood samples for CTC detection according to the wishes of patients.
  Patients underwent contrast-enhanced thoracoabdominal and pelvic Computer Tomography(CT) at baseline and every 6 weeks after enrollment. Patients with stable or remission after 2 to 6 cycles of combined treatment can reduce the evaluation frequency to once every 12 weeks during the maintenance treatment period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment of HER-2 Negative MSS Advanced Gastric (Experimental): Sintilimab Plus Apatinib and Chemotherapy in Patients with Previously Untreated HER-2 negative MSS Advanced or Metastatic GC or GEJ Cancer
  Interventions: Drug: Sintilimab 200 mg, intravenously (IV) every 3 weeks(Q3W)

INTERVENTIONS:
Drug: Sintilimab 200 mg, intravenously (IV) every 3 weeks(Q3W) — for 2-6 cycles followed by Sindilizumab plus Tegafur gimeracil oteracil potassium capsules.
  Other Names: Apatinib 250 mg twice daily (BID) by continous oral adminstration for 14 days, followed by a recovery period of 7 days;; Tegafur gimeracil oteracil potassium capsules twice daily (BID) by continous oral adminstration for 14 days, every 3 weeks(Q3W); Oxaliplatin 85 mg/m^2, IV every 3 weeks(Q3W)

SUMMARY:
To evaluate the efficacy and safety of Sintilimab combined with apatinib and chemotherapy as First-line or second-line Therapy in Treatment of HER-2 negative MSS Advanced or Metastatic GC or GEJ Cancer. At the same time, the correlation between tissue programmed death ligand-1(PD-L1) expression and blood circulating tumor cell(CTC) counts and the efficacy of immune combination therapy was also explored.

DETAILED DESCRIPTION:
Participants receive Sintilizumab 200 mg, intravenously (IV) every 3 weeks(Q3W);plus Apatinib 250 mg twice daily (BID) by continous oral adminstration for 14 days, followed by a recovery period of 7 days; plus Tegafur gimeracil oteracil potassium capsules (40mg for body surface area < 1.25/m^2, 50mg/m^2 for body surface area 1.25-1.5m^2, 60mg for body surface area > 1.5/m^2) BID by continous oral adminstration for 14 days, followed by a recovery period of 7 days, plus Oxaliplatin 85 mg/m^2, IV Q3W; for 4-6 cycles followed by Cindilizumab plus Tegafur gimeracil oteracil potassium capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with inoperable advanced, recurrent or metastatic gastric and gastroesophageal junction adenocarcinoma confirmed by histology, and HER-2 negative by immunohistochemistry. HER-2 negative was defined as immunohistochemistry 0-1 + or 2 + but fish results were negative.
2. According to recist1 1 measurement standard at least one or more target lesions can be measured.
3. Patients with microsatellite stability (MSS type) or normal mismatch repair protein (PMMR) confirmed by immunohistochemistry or second-generation sequencing..
4. Aged 18-75.
5. The performance status of the Eastern Cooperative Oncology Group (ECOG) is 0-1 points.
6. Life expectancy is more than 3 months.
7. The blood routine examination was basically normal within 1 week before enrollment (taking the normal value in the laboratory of each research center as the standard). The white blood cell count (WBC) ≥ 2.5 × 10^9 / L or neutrophil count (ANC) ≥ 1.5 × 10^9/L; Platelet count (PLT) ≥ 100 × 10^9/L； Hemoglobin ≥ 9.0 g / dl. Patients can receive blood transfusion or erythropoietin treatment to meet this standard.
8. The liver and kidney function, nail function and coagulation function were basically normal within 1 week before enrollment (based on the normal values in the laboratories of each research center). Total bilirubin (TBIL) ≤ 1.5 × Upper limit of normal value (ULN); alanine aminotransferase (SGPT / ALT) ≤ 2.5 × ULN (patients with liver metastasis) ≤ 5 × ULN);Aspartate aminotransferase (SGOT / AST) ≤ 2.5 × ULN (patients with liver metastasis) ≤ 5 × ULN);Creatinine clearance rate (CCR) ≥ 60 ml / min; Urinary protein < 2 +; If urinary protein ≥ 2 +, 24-hour urinary protein must be ≤ 1g; Thyroid stimulating hormone (TSH) ≤ upper limit of normal value (ULN); in case of abnormality, T3 and T4 levels shall be measured; if T3 and T4 levels are normal, they can be selected. International normalized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN。
9. The patient is willing and able to comply with the provisions of the study protocol during the study.
10. Before entering the study, during the study and within 6 months after the end of treatment, patients with fertility must take effective contraceptive measures (hormone or barrier contraception; abstinence).
11. The subject agreed not to participate in another intervention study when receiving the study drug in this study. Subjects ended the last study for more than 1 month.
12. Subjects who have received adjuvant or neoadjuvant therapy (including chemotherapy, radiotherapy or chemoradiotherapy) of GC / GEJ must complete the last dose of treatment at least 6 months before the first study treatment. Palliative radiotherapy is allowed, but it must be completed 2 weeks before the start of study treatment.

Exclusion Criteria:

1. Patients who have received chemotherapy, radiotherapy or biological therapy within two weeks. Received any investigational drug within 4 weeks before the start of study treatment.
2. Pregnant or lactating women; women with fertility have a positive pregnancy test or no pregnancy test at the time of screening.
3. Severe / uncontrolled intermittent disease / infection.
4. Obvious cardiovascular disease (history of congestive heart failure > NYHA class II, unstable angina pectoris or myocardial infarction, unstable angina pectoris or myocardial infarction, or severe arrhythmia in the past six months).
5. History or evidence of hereditary bleeding syndrome or coagulation disease with bleeding risk, history of thrombotic disease and active gastrointestinal bleeding.
6. There have been arterial thromboembolism events in the past 6 months, including transient ischemic attack and cerebrovascular accident.
7. Patients with previous malignant tumors, unless the previous malignant tumors have been diagnosed and treated for more than 5 years, and there is no evidence of recurrence.
8. The subjects have known human immunodeficiency virus (HIV) infection or known positive detection history of active hepatitis B (positive HBsAg) or hepatitis C infection. The subjects with HBsAg negative but HBC AB positive will be tested for HBV DNA replication. If it is greater than the minimum copy number of HBV DNA, the subjects will be excluded. The subjects with seropositive but hepatitis C virus The subjects with negative replication results of (HCV) RNA test are eligible for inclusion.
9. Patients with neuropathy > grade 3 at screening.
10. Patients with QTc > 500msec during screening.
11. Patients with meningeal disease and no other measurable brain metastasis were excluded.
12. Have received bevacizumab, sorafenib, sunitinib or other VEGF pathway targeted therapy.
13. Have a history of severe hemoptysis.
14. Having a mental illness or social situation can hinder study compliance.
15. A severe nonunion wound, ulcer, or bone fracture.
16. Major surgery, open biopsy or major trauma within 28 days before enrollment, and minor surgery within 7 days before enrollment.
17. Have a history of allergic reaction to compounds similar to the chemical composition of the study drug.
18. Take chronic daily aspirin (> 325 mg / day), dipyridamole, ticlopidine, clopidogrel, cilostazol, non steroidal anti-inflammatory drugs and other drugs known to inhibit platelet function.
19. Recent formal antihypertensive treatment still failed to control hypertension (systolic blood pressure greater than 140mmHg and diastolic blood pressure greater than 90mmHg), and the patients had obvious symptoms of hypertension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 31 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 36 months
  per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 36 months
  per RECIST 1.1
Disease Control Rate (DCR) | 36 months
  per RECIST 1.1
Duration of Response (DoR) | 36 months
  per RECIST 1.1
Adverse events (AEs) | 36 months
  Number of Subjects with treatment-related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Qinghai University, Xining, Qinghai, China